CLINICAL TRIAL: NCT06371846
Title: Comparative Study of the Surface and Endocavitary Signals of Cardiac Pacing System Analyzers With Respect to the Conventional Polygraphy Systems Signals During Implantation of Conduction System Pacing Devices
Brief Title: Comparative Study of the Surface Electrocardiogram Signals During the Implantation of Conduction System Pacing Devices
Status: Recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: 2023 /10850/I
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Conduction Disorder; Pacemaker DDD
Keywords: Conduction Pacing System; Program System Analyzers
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort one: This was a non-randomized, prospective multicentric study. From july 2023 to may 2024 consecutive patients over 18 years of age who underwent a LBBAP system as first intention, were enrolled from five participating hospitals. Baseline characteristics including demography, pacing indication, basal QRS and left ventricular ejection fraction were collected. For the implantation procedure analysis, total procedural time, total fluoroscopy time, total radiation dosage, pacing electrocardiogram parameters including the paced QRS morphology and duration, V6 R wave peak time (V6-RWPT), and changes between selective and non-selective LBBP were recorded, as well as the pacing lead parameters including R-wave amplitude, threshold and impedance with unipolar and bipolar configurations. First 24hs complications were all documented.
  Interventions: Other: Selected signals from Pacing System Analyzers

INTERVENTIONS:
Other: Selected signals from Pacing System Analyzers — Comparative observational, prospective, multicenter study between the signals obtained by PSA vs MPS of consecutive patients who underwent a LBBAP strategy as first intention.

SUMMARY:
Introduction and objectives: Left bundle branch area pacing (LBBAP), is a novel modality of physiologic pacing that requires an adequate assessment of the endocardium as well as the body-surface electrocardiographic signals for a successful pacing-lead implantation. The objective of the study consist of assessing if LBBAP criteria, specifically septal and left bundle branch pacing (LBBP) criteria, can be satisfactory measured using the signals resulting from different cardiac pacing analyzers (PSAs) by comparing them to the 'conventional' signals obtained from multichannel polygraph systems (MPSs) during the implantation procedure.

Methods: Comparative observational, prospective, multicenter study between the signals obtained by PSA vs MPS of consecutive patients who underwent a LBBAP strategy as first intention.

DETAILED DESCRIPTION:
METHODS All participants will provide written informed consent before undergoing the procedure. The study was approved by the Institutional Review Board of Hospital del Mar (Barcelona) and complied with the declaration of Helsinki.

Study protocol and data collection This was a non-randomized, prospective multicentric study. From july 2023 to may 2024 consecutive patients over 18 years of age who will undergo a LBBAP system as first intention, will be enrolled from five participating hospitals. Baseline characteristics including demography, pacing indication, basal QRS and left ventricular ejection fraction will be collected. For the implantation procedure analysis, total procedural time, total fluoroscopy time, total radiation dosage, pacing electrocardiogram parameters including the paced QRS morphology and duration, V6 R wave peak time (V6-RWPT), and changes between selective and non-selective LBBP will be recorded, as well as the pacing lead parameters including R-wave amplitude, threshold and impedance with unipolar and bipolar configurations. First 24hs complications will be all documented.

In a prephase of the study, a comparison between MPS and PSA surface signals, was performed. Medtronic and Biotronik PSAs' use a four-leads monitoring system, three of them detecting bipolar signals. The Right Arm (RA) lead was placed at the back of the patient, at the level of the heart, to diminish the distance between leads and generating two 'pseudomonopolar' signals together with the two other leads, (Left Arm (LA) and Left Foot (LF)) placed at "V1" and "V6" standard positions ("modified" leads position). Boston Scientific (BSC) and Abbott PSAs use a five-leads monitoring system, one of them (V1 lead) capable of detecting a monopolar signal. In this case, the V1 lead was placed at the standard "V1" position and the LA lead was moved to the "V6" position ("modified" lead position). The similarities on the QRS morphology compared to the MPS were confirmed in all PSAs.

Implantation procedure All patients received standard medical treatment according to their clinical conditions and underwent the LBBAP implantation in accordance with the standardized pacemaker implantation technique. Bipolar electrograms were filtered through a bandpass of 30-500 Hertz (Hz) and recorded on a MPS at a speed of 100milimeter/second (mm/s) and a gain of 0.1 miliVolt/centimeter (mV/cm). Before the implantation procedure, the PSA-leads will be placed as previously described. Signals will be optimized and displayed in each PSA screen at a speed range between [50-100] mm/sec and at gain of 0.05 mV/mm. The basal QRS morphology and duration corresponding to 'V1' and 'V6' PSA-leads will be compared to those of the MSP, to assess the correct position of the electrodes. In case of detecting a QRS morphology and/or duration on the PSA significantly different from the MSP (more than 2 deflections in opposite directions or a difference in QRS duration > 10 msec), repositioning of the leads wil be suggested to obtain a similar QRS morphology and duration between both recording systems. The sheath as well as the pacing-lead characteristics and final position (LVSP vs LBBP) will be left at operator's discretion.

Left bundle branch (LBB) capture was defined in the presence of a paced QRS with right bundle branch block (RBBB) morphology in V1 (initial r wave in lead V1) and at least one of the following criteria:

1. V6-RWPT < 80 msec.
2. V1-V6 inter-peak interval > 33 msec.
3. QRS transition from non-selective left bundle branch pacing (NS-LBBP) to selective left bundle branch pacing (S-LBBP) or NS-LBBP to left ventricular septal pacing (LVSP) during pacing threshold.
4. Sudden increase of V6-RWPT > 15 msec because of reducing pacing output.
5. Left bundle potential-V6RWPT = stim-V6RWPT (±10 msec). For patients without initial r wave in V1, LBBP will be considered in the presence of QRS transition during pacing. LVSP will be defined by a paced QRS showing a typical terminal R-wave in V1, anatomical position of the lead in the left ventricular septum documented by fluoroscopy and not fulfilling the additional criteria previously described for LBBP.

During the implant procedure, initial septal unipolar pacing will be performed looking for an "W" morphology in V1 in the mid-septal area, and the last recommendations of international guidelines will be followed for placing the lead. Briefly, when the selected initial position at operator's discretion is fulfilled, the lead is deployed using rapid turns and lead depth within the septum is assessed using pacing QRS morphology, pacing impedance, unfiltered electrogram amplitude from lead tip, or using contrast through the sheath. The objective of the study is to validate and compare the criteria for the LBBAP in both recording systems. Specifically, paced QRS in V1 and V6, V6-RWPT, V1-V6 inter-peak interval, abrupt Δ V6-RWPT > 15 msec at decremental pacing output and QRS transitions between non-selective and selective capture of the conduction system during pacing were measured and confirmed in both, the PSA and the MSP, to assess the final lead position. Endocavitary signals from the lead tip will be evaluated and measured to detect congruent pre-ventricular signals from the conduction system as well.

Monitoring and discharge Patients will be in-hospital for a period of 24 hours. Before discharge, all patients will undergo a 12-lead electrocardiogram, an X-ray in postero-anterior and lateral views, as well as clinical monitoring to rule out acute complications.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age who underwent a LBBAP system as first intention.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who underwent a left bundle branch area pacing system as first intention
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Similarity of signals between multichannel recording system and Pacing System Analyzers | First 24 hours
  To describe the similarity of signals between multichannel recording system and Pacing System Analyzers

SECONDARY OUTCOMES:
Security | First 24 hours
  To describe the incidence of pneumothorax, bleeding, electrode perforation and/or cardiac tamponade, lead dislodgement or infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Jiménez López, MD, Principal Investigator — Cardiac Electrophysiologist
Locations (1):
- Jesus Jiménez López, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Each researcher only have their own available data except for the main researcher, who have all data centers, but without any identity of the patient.